CLINICAL TRIAL: NCT03329521
Title: Multicomponent Intervention to Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD) in Patients With Chronic Kidney Disease: A Pragmatic, Registry-based, Cluster-Randomized Clinical Trial
Brief Title: Enhance Access to Kidney Transplantation and Living Kidney Donation
Acronym: EnAKT LKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Institute for Clinical Evaluative Sciences (ICES) (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Renal Network (part of Ontario Health) (Unknown); Trillium Gift of Life Network (part of Ontario Health) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R-17-088
Record Dates: First submitted 2017-09-29; First posted 2017-11-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Kidney Diseases; Kidney Failure; End Stage Renal Disease
Keywords: Cluster Randomized Controlled Trial; Kidney Transplant; Living Kidney Donation; Kidney Disease
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent intervention (Experimental): A multicomponent intervention will be provided at chronic kidney disease (CKD) programs.
  Interventions: Other: Multicomponent intervention
- Usual Care (No Intervention): CKD programs will continue to support access to kidney transplantation and living kidney donation as they usually do for CKD patients.

INTERVENTIONS:
Other: Multicomponent intervention — Patients in 13 of the 26 CKD programs will receive a multicomponent intervention or usual care. The intervention has four main components: (1) support for local quality improvement teams and administrative needs; (2) tailored education and resources for staff, patients, and living kidney donor candidates; (3) support from kidney transplant recipients and living kidney donors; and (4) program-level performance reports and oversight by program leaders.
  Arms: Multicomponent intervention

SUMMARY:
Compared to dialysis, kidney transplantation is associated with improved survival, better quality of life and substantial cost savings to healthcare systems. Despite these advantages, many individuals with kidney failure will never receive a kidney transplant. A multicomponent intervention (vs. usual care) provided in chronic kidney disease (CKD) programs located in Ontario, Canada was developed to determine if it can enable more patients with no recorded contraindications to kidney transplant to complete more steps towards receiving a kidney transplant. These CKD programs provide care to individuals with CKD (including patients approaching the need for dialysis and patients receiving dialysis). The intervention has four main components: (1) support for local quality improvement teams and administrative needs; (2) tailored education and resources for staff, patients, and living kidney donor candidates; (3) support from kidney transplant recipients and living kidney donors (i.e. Transplant Ambassador Program); and (4) program-level performance reports and oversight by program leaders. The Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD) trial will provide high-quality evidence on whether a multicomponent intervention helps patients complete more steps towards receiving a kidney transplant.

DETAILED DESCRIPTION:
1. Statement of the health problem or issue: Compared with dialysis, a kidney transplant offers patients a better quality of life and many gain 10 or more years of life expectancy. A transplant also costs the healthcare system less-over a five-year period. Living donor transplants offer further advantages, including superior graft and patient survival compared with deceased donor transplants. Unfortunately, many patients with kidney failure who would benefit from a transplant will never receive one. There is a chronic shortage of organs from deceased donors, and in Canada, the rate of living donor kidney transplantation has stagnated. In addition to the shortage of transplantable kidneys, several other barriers impede patient access to transplantation.
2. Objective of your project: To determine if a multicomponent intervention provided in chronic kidney disease (CKD) programs (vs. usual care) enables more patients with no recorded contraindications to kidney transplant to complete more steps towards receiving a kidney transplant.
3. How will you undertake your work? We will conduct a pragmatic two-arm, parallel-group, open-label, registry-based, cluster-randomized, superiority, clinical trial-the Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD) trial. Our study will include the 26 chronic kidney disease (CKD) programs in Ontario, Canada which are expected to care for over 10,000 adult patients with CKD (including patients approaching the need for dialysis and patients receiving dialysis) with no recorded contraindications to a kidney transplant during the trial. Patients in 13 of the 26 CKD programs will receive a multicomponent intervention or usual care. The intervention has four main components: (1) support for local quality improvement teams and administrative needs; (2) tailored education and resources for staff, patients, and living kidney donor candidates; (3) support from kidney transplant recipients and living kidney donors; and (4) program-level performance reports and oversight by program leaders. Patients in the other 13 programs will receive usual care and will continue to receive support in accessing kidney transplantation and living kidney donation as usual.
4. What is unique/innovative about your project? An investigator usually needs to study a large number of patients in a clinical trial to reliably understand the effects of an intervention. Normally, a study with 10,000 patients would cost more than $10 million dollars to conduct; however, this study will provide a reliable answer to the question being asked and can be done at a fraction of the cost. This is because we will use data routinely collected by the healthcare system. The investigator will be able to analyze these healthcare data at the end of the study. This means that the study will cost less than a traditional clinical trial. Also unique to this trial, is that that the intervention was embedded and delivered in routine care.

   This pragmatic trial includes all CKD programs in the province of Ontario. By including patients from a variety of backgrounds, the results of the trial should be broadly generalizable.
5. What is the impact of the proposed research? The EnAKT LKD trial will provide high-quality evidence on whether a multicomponent intervention helps patients complete more steps towards receiving a kidney transplant. This is important as compared to dialysis, kidney transplant offers patients a better quality of life and many gain 10 or more years of life expectancy. A transplant also costs the healthcare system less. If our intervention is successful, more transplants may ultimately be performed and result in improved survival and a better quality of life for patients with CKD. Kidney transplantation achieves the triple aim in healthcare: better outcomes, better experience of care, and lower costs.

ELIGIBILITY:
This is a pragmatic, two-arm, parallel-group, open-label, registry-based cluster randomized, superiority, clinical trial with eligibility criteria detailed below.

Inclusion Criteria:

* All 26 chronic kidney disease (CKD) programs in Ontario. These programs provide care for all chronic dialysis patients in the province. Each CKD program also provides a multi-care kidney clinic for patients with advanced CKD who are approaching the need for dialysis.

Exclusion Criteria:

* None. Including all Ontario CKD programs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Completing key steps toward receiving a kidney transplant | 4.17 years
  The primary outcome is completing key steps toward receiving a kidney transplant, where up to 4 unique steps per patient will be considered: (1) patient referred to a transplant center for evaluation, (2) a potential living kidney donor begins their evaluation at a transplant center to donate a kidney to the patient, (3) patient added to the deceased donor transplant wait list, and (4) patient receives a kidney transplant from a living or deceased donor.

SECONDARY OUTCOMES:
A potential living kidney donor begins their evaluation at a transplant center to donate a kidney to the patient and/or a patient receives a living donor transplant. | 4.17 years
  Given that the average wait time for a deceased donor kidney transplant is five years on average in Ontario, our intervention is likely to have only a small impact on the rate of deceased donor kidney transplants. For this reason, we have pre-specified five secondary outcomes to examine the impact of our intervention on living kidney donor transplant activity.
Time to first occurrence of a potential living kidney donor beginning their evaluation at a transplant center to donate a kidney to the patient. | 4.17 years
  Secondary outcome selected to understand living kidney donor transplant activity.
A transplant center receives a patient's complete referral package from a chronic kidney disease program and at least one potential living kidney donor begins their evaluation at a transplant center to donate a kidney to the patient. | 4.17 years
  Secondary outcome selected to understand living kidney donor transplant activity.
A patient receives a living donor kidney transplant | 4.17 years
  Secondary outcome selected to understand living kidney donor transplant activity.
A patient receives a pre-emptive living donor kidney transplant (restricted to patients who were not receiving dialysis when they entered the trial and not on dialysis at the time of transplant). | 4.17 years
  Secondary outcome selected to understand living kidney donor transplant activity.

OTHER OUTCOMES:
Rate of deceased donor kidney transplant | 4.17 years
  Rate of deceased donor kidney transplant censoring at receipt of a living donor kidney transplant and at the censoring events included in the main trial analysis (i.e., emigration, trial end date [December 31, 2021], death, evidence of recovered kidney function, or on the date a recorded contraindication to transplant occurs [with the exception of age >75]).
Average number of months from the date of dialysis initiation (i.e. trial entry) to the date of referral | 4.17 years
  This outcome is assessed in patients receiving maintenance dialysis who were referred to a transplant centre.
Rate of living kidney donor transplants | 4.17 years
  This outcome is assessed in patients waitlisted for a deceased donor kidney transplant and censored at receipt of a deceased donor kidney transplant and at the censoring events included in the main trial analysis (i.e., emigration, trial end date [December 31, 2021], death, evidence of recovered kidney function, or on the date a recorded contraindication to transplant occurs [with the exception of age >75]).
Proportion of pre-emptive transplants | 4.17 years
  This outcome is assessed in recipients of a living kidney donor transplant and restricted to patients who were not receiving dialysis when they entered the trial and not on dialysis at the time of transplant.
Average number of months from the date of referral to a transplant center to the date the first living donor candidate contacts the transplant centre for the intended recipient | 4.17 years
  This outcome is assessed in recipients of a living kidney donor transplant.
Average number of months from the date of referral to a transplant center to date of the transplant surgery | 4.17 years
  This outcome is assessed in recipients of a living or deceased donor kidney transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, MD, PhD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
While data sharing agreements prohibit ICES from making the data publicly available, access may be granted to those who meet prespecified criteria for confidential access, available at www.ices.on.ca/DAS. The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the programs may rely upon coding templates or macros that are unique to ICES.

REFERENCES:
- [Background] Yohanna S, Naylor KL, Mucsi I, McKenzie S, Belenko D, Blake PG, Coghlan C, Dixon SN, Elliott L, Getchell L, Ki V, Nesrallah G, Patzer RE, Presseau J, Reich M, Sontrop JM, Treleaven D, Waterman AD, Zaltzman J, Garg AX on behalf of the EnAKT LKD investigators. A Quality Improvement Intervention to Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD) in Patients With Chronic Kidney Disease: Clinical Research Protocol of a Cluster-Randomized Clinical Trial. Can J Kidney Health Dis. 2021 Apr 15;8:doi:10.1177/2054358121997266.
- [Background] Naylor KL, McKenzie SQ, Garg AX, Yohanna S, Sontrop JM. Partnering with Patients to Enhance Access to Kidney Transplantation and Living Kidney Donation. Healthc Q. 2022 Apr;24(SP):69-73. doi: 10.12927/hcq.2022.26771. PMID 35467514
- [Background] Dixon SN, Naylor KL, Yohanna S, McKenzie S, Belenko D, Blake PG, Coghlan C, Cooper R, Elliott L, Getchell L, Ki V, Mucsi I, Nesrallah G, Patzer RE, Presseau J, Reich M, Sontrop JM, Treleaven D, Waterman AD, Zaltzman J, Garg AX. Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD): Statistical Analysis Plan of a Registry-Based, Cluster-Randomized Clinical Trial. Can J Kidney Health Dis. 2022 Nov 22;9:20543581221131201. doi: 10.1177/20543581221131201. eCollection 2022. PMID 36438439
- [Background] Yohanna S, Wilson M, Naylor KL, Garg AX, Sontrop JM, Belenko D, Elliott L, McKenzie S, Macanovic S, Mucsi I, Patzer R, Voronin I, Lui I, Blake PG, Waterman AD, Treleaven D, Presseau J. Protocol for a Process Evaluation of the Quality Improvement Intervention to Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD) Cluster-Randomized Clinical Trial. Can J Kidney Health Dis. 2022 Mar 19;9:20543581221084502. doi: 10.1177/20543581221084502. eCollection 2022. PMID 35340770
- [Background] Garg AX, Yohanna S, Naylor KL, McKenzie SQ, Mucsi I, Dixon SN, Luo B, Sontrop JM, Beaucage M, Belenko D, Coghlan C, Cooper R, Elliott L, Getchell L, Heale E, Ki V, Nesrallah G, Patzer RE, Presseau J, Reich M, Treleaven D, Wang C, Waterman AD, Zaltzman J, Blake PG. Effect of a Novel Multicomponent Intervention to Improve Patient Access to Kidney Transplant and Living Kidney Donation: The EnAKT LKD Cluster Randomized Clinical Trial. JAMA Intern Med. 2023 Dec 1;183(12):1366-1375. doi: 10.1001/jamainternmed.2023.5802. PMID 37922156
- [Derived] Yohanna S, Wilson M, Naylor KL, Garg AX, Sontrop JM, Mucsi I, Belenko D, Dixon SN, Blake PG, Cooper R, Elliott L, Heale E, Macanovic S, Patzer R, Waterman AD, Treleaven D, Coghlan C, Reich M, McKenzie S, Presseau J. Process Evaluation Alongside a Cluster-Randomized Trial of a Multicomponent Intervention Designed to Improve Patient Access to Kidney Transplantation. Can J Kidney Health Dis. 2025 Mar 17;12:20543581251323959. doi: 10.1177/20543581251323959. eCollection 2025. PMID 40104388
- [Derived] Yohanna S, Naylor KL, Mucsi I, McKenzie S, Belenko D, Blake PG, Coghlan C, Dixon SN, Elliott L, Getchell L, Ki V, Nesrallah G, Patzer RE, Presseau J, Reich M, Sontrop JM, Treleaven D, Waterman AD, Zaltzman J, Garg AX. A Quality Improvement Intervention to Enhance Access to Kidney Transplantation and Living Kidney Donation (EnAKT LKD) in Patients With Chronic Kidney Disease: Clinical Research Protocol of a Cluster-Randomized Clinical Trial. Can J Kidney Health Dis. 2021 Apr 15;8:2054358121997266. doi: 10.1177/2054358121997266. eCollection 2021. PMID 33948191

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT03329521/Prot_SAP_002.pdf